CLINICAL TRIAL: NCT05041088
Title: ProdromeNeuro: A Phase I Study of Omega 3 Oil Nutritional Supplementation for Aging-Related Cognitive Decline
Brief Title: Omega 3 Oil: Aging-Related Cognitive Decline
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neurological Associates of West Los Angeles (Other)
Collaborators: Prodrome Sciences Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Plasmalogen2.0
Record Dates: First submitted 2021-08-30; First posted 2021-09-10 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Aging Related Cognitive Decline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (ALL participants) (Experimental): This group will be taking plamalogen supplement (ProdromeNeuro) and be followed through the study with neuropsychological testing, serology, and follow up MRI data. They will be administered 2mL per day for 6 months
  Interventions: Dietary Supplement: ProdromeNeuro Plasmalogen

INTERVENTIONS:
Dietary Supplement: ProdromeNeuro Plasmalogen — The product being investigated in this study is the ProdromeNeuro Omega 3 oil nutritional supplement. This product contains naturally occurring fatty acids in higher concentrations than similar products that are commercially available. The purpose of this research study is to better understand the effects of ProdromeNeuro Omega-3 nutritional supplementation among participants with age-related cognitive decline.

SUMMARY:
Aging-related cognitive decline may be affected by brain cholesterol and the health of cell membranes. Certain nutritional supplements have been proposed to support membrane health, and there is increasing interest in plasmalogens and Omega-3 derived oil supplements to support brain health among older adults. Plasmalogens are compounds found in neural cell membranes that are connected to cholesterol processing. Neural cells that have low plasmalogens have shown an inability to process cholesterol properly. Recent research suggests that abnormalities in cholesterol processing and low levels of plasmalogen may play a role in age-related cognitive decline.

The product being investigated in this study is the ProdromeNeuro Omega 3 oil nutritional supplement. This product contains naturally occurring fatty acids in higher concentrations than similar products that are commercially available. The purpose of this research study is to better understand the effects of ProdromeNeuro Omega-3 nutritional supplementation among participants with age-related cognitive decline. It is hoped that taking this product over the course of 4 months will result in improved plasmalogen levels, brain connectivity seen on advanced brain imaging, as well as improved cognitive assessment measurements.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a degenerative process
* Clinical Dementia Rating (CDR) score indicating mild cognitive impairment (CDR = 0.5), mild dementia (CDR = 1) through moderate dementia (CDR = 2)

Exclusion Criteria:

* Subjects unable to give informed assent
* Cognitive decline clearly related to an acute illness
* Advanced terminal illness
* Any active cancer or chemotherapy
* Any other neoplastic illness or illness characterized by neovascularity or angiopathy
* Subjects previously taking plasmalogen supplementation prior to study enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
Change in ProdromeScan Blood Test | Change monitored from baseline to 6 month time point (also assessed for change at the end of each month is this time period)
  serological testing kit for plasmalogen levels

SECONDARY OUTCOMES:
Change in 9-Hole Pegboard Task (9-HPT) | Change monitored from baseline to 6 month time point (also assessed for change at the end of each month is this time period)
  A validated assessment for fine motor skills, the 9-HPT involves having a participant move 9 pegs individually from starting position to 9 separate peg-holes, as quickly as possible, and to immediately return the 9 pegs to the starting position upon filling the final peg-hole. This is performed separately for each hand. The score is the time (seconds/milliseconds) that it takes to complete the task, recorded separately for dominant and non-dominant hands. The minimum detectable change is 2.6 seconds for the dominant hand and 1.3 seconds for the non-dominant hand.
Change in Montreal Cognitive Assessment (MoCA) | Change monitored from baseline to 6 month time point (also assessed for change at the end of each month is this time period)
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.
Change in Timed 25-foot Walk Test (T25-FW) | Change monitored from baseline to 6 month time point (also assessed for change at the end of each month is this time period)
  The T25FW is a clinical tool that evaluates patients for quantitative mobility and leg function performance test in a timed, 25-foot walk. Scoring for this task is the average number of steps (from first step to the first heel-strike after the finish line) and time taken (seconds/milliseconds) of two trials. Minimally clinically important difference (MCID) is 20% improvement in time taken and/or number of steps taken to complete.
Change in Timed 25-foot Walk Test Steps (T25-FW) | Change monitored from baseline to 6 month time point (also assessed for change at the end of each month is this time period)
  The T25FW is a clinical tool that evaluates patients for quantitative mobility and leg function performance test in a timed, 25-foot walk. Scoring for this task is the average number of steps (from first step to the first heel-strike after the finish line) of two trials. Minimally clinically important difference (MCID) is 20% improvement in number of steps taken to complete.
Change in 30-Second Sit Stand (30CST) | Change monitored from baseline to 6 month time point (also assessed for change at the end of each month is this time period)
  The 30-second chair stand involves recording the number of times that a person can complete a full stand in 30 seconds. This measure assesses functional lower extremity strength in older adults. The participant is instructed to complete as many full stands as possible within 30 seconds, starting in a seated position in the middle of an armless chair. The participant is instructed to fully sit between each stand. The tester silently counts the completion of each correct stand, and the score is the total number of stands within 30 seconds. The minimum clinically important difference (MCID) is 2 full stands per 30 second testing.
Change in Quick Dementia Rating Scale (QDRS) used to calculate a Clinical Dementia Rating (CDR) scale | Change monitored from baseline to 6 month time point (also assessed for change at the end of each month is this time period)
  The Quick Dementia Rating Scale (QDRS) is an interview-based tool administered by study officials to participants' caregivers used to obtain observations from a consistent source. The QDRS form consists of 10 categorical questions (5 cognitive, 5 functional), each with 5 detailed options depicting the level of impairment as either 0 (normal), 0.5 (mild/inconsistent impairment), 1 (mild/consistent impairment), 2 (moderate impairment), or 3 (severe impairment). Based on the conversion table outlined in Dr. James Galvin's research (2015), total QDRS scores were converted to Clinical Dementia Rating (CDR) scale levels ranging from 0 (normal aging), 0.5 (mild cognitive impairment), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia).
Global Rating of Change (GRC) | Assessed at 6 month time point (reflecting on the study)
  GThe GRC consists of a single likert-scale ranging from "-5" (very much worse) to "0" (neutral/no change) to "5" (very much better). The GRC is obtained in an interview format to assess a patient's perceived change in status following a treatment. A score that is at least 2 or greater is considered to indicate clinically significant change.
Change in Timed 25-foot Walk Test Speed (T25-FW) | Change monitored from baseline to 6 month time point (also assessed for change at the end of each month is this time period)
  The T25FW is a clinical tool that evaluates patients for quantitative mobility and leg function performance test in a timed, 25-foot walk. Scoring for this task is the average time to complete walk (in seconds/milliseconds) (from first step to the first heel-strike after the finish line) of two trials. Minimally clinically important difference (MCID) is 20% improvement in time taken to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Kennedy Mahdavi, BS, Study Director — Neurological Associates; Sheldon Jordan, MD, Principal Investigator — Neurological Associates

IPD SHARING:
Plan to Share IPD: No